CLINICAL TRIAL: NCT04653688
Title: A Prospective Study on Markers of Disease Progression and Gait Within the Parkinsonian Population
Brief Title: Markers of Disease Progression and Gait Within the Parkinsonian Population
Acronym: Gait'N'Park
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: H. Lundbeck A/S (Industry); France Parkinson Association (Other); Vaincre Parkinson (Unknown); FeetMe (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2019_64; 2020-A01998-31 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-10-06; First posted 2020-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Gait disorders; On-OFF detection; FOG detection; Quality of life; personalize medicine; telemedicine
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation | interventions — ioflupane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinsonian syndromes patients (Experimental)
  Interventions: Device: The FeetMe® Evaluation; Device: the PKG® Watch,; Radiation: MRI; Radiation: DaTSCAN
- healthy subjects (Sham Comparator)
  Interventions: Device: The FeetMe® Evaluation; Radiation: MRI

INTERVENTIONS:
Device: The FeetMe® Evaluation — The FeetMe® Evaluation device is a medical device (class Im CE 0459) for ambulatory gait analysis, consisting of a pair of connected insoles and an Android mobile application.
Device: the PKG® Watch, — The PKG® provides continuous, objective, ambulatory assessment of the treatable and disabling symptoms of Parkinson's disease including tremor, bradykinesia and dyskinesia. The PKG® system consists of a wrist-worn movement recording device known as the PKG® Watch,
  Arms: Parkinsonian syndromes patients
Radiation: MRI — * an anatomical 3D T1-weigthed gradient-echo sequence (1mm isotropic):
  * anatomical registration
  * automated segmentation
  * volumetric
  * texture analysis
Radiation: DaTSCAN — * quantify nigrostriatal dopaminergic depletion
  * correlate its impact on the type and severity of gait disorders in Parkinson's disease.
  Arms: Parkinsonian syndromes patients

SUMMARY:
The aim of the project is to evaluate disease progression of patients with Parkinsonian syndrome of various severity through regular home-based gait parameters analysis.

We identified several steps in this project:

1. Acquisition of gait data in 120 patients with Parkinsonism at different stages in hospital and ecological condition (during 10 days at home), in a repetitive manner:

   1. 30 Early PD patients, before 3 years of disease duration (MDS criteria, 2018)
   2. 30 PD patients with motor fluctuations (5 to 8 years of disease duration) (MDS criteria, 2018)
   3. 30 PD patients with FoG (10 years of disease duration) (MDS criteria, 2018)
   4. 30 patients with MSA (less than 5 years after the first symptom)
2. Control groups will be composed by 30 healthy volunteers Correlation analysis with clinical measurements and biomarkers, namely blood biomarkers for neurodegeneration (4HN, NFLT …) and multimodal MRI repeated assessments (Iron overload, inflammation and degeneration) and genetic panel for common haplotypes involved in Parkinsonism.

ELIGIBILITY:
Inclusion Criteria:

PD Patients:

* Age: from 40 to 80 years
* Absence of intercurrent pathology that may interfere with the purpose of the study (rheumatologic or orthopedic condition, cardiac, severe pulmonary disease that may limit the perimeter of walking)

Each group will be composed of:

* 30 PD with a disease duration < 3 years
* 30 PD with a disease duration between 5 to 8 years
* 30 PD with a disease duration > 10 years MSA Patients
* Age > 30 years old
* < 5 years of disease duration
* deemed by the physicians to be able to walk at 1 year

Healthy subjects

• Similar age and sex distribution

For all

* Absence of intercurrent pathology that may interfere with the purpose of the study (rheumatologic or orthopedic condition, cardiac, severe pulmonary disease that may limit the perimeter of walking)
* Absence of cognitive disorders (MoCA> 24/30 according to the MDS criteria)
* Stable treatment for at least 2 weeks before inclusion
* Ability to walk at least 100 meters
* Have an affiliation to the social security or equivalent
* Have signed an informed consent

Exclusion Criteria:

* STN DBS for PD patients
* Intraduodeno-jejunal levodopa infusion (duodopa)
* Inability to walk without aid (walker or walking stick)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Changes of 95th percentile of home gait velocity (assessed during 10 days with FeetMe® Insoles) at 48 weeks versus baseline in Parkinsonian syndrome patient subgroups and in a control group. | at 48 weeks

SECONDARY OUTCOMES:
Changes of 95th percentile of home gait velocity (assessed during 10 days with FeetMe® Insoles) at 12 weeks (MSA subgroup only) and 24 weeks versus baseline in Parkinsonian syndrome patient subgroups | at baseline at 12weeks, at 24 weeks and 48 weeks
Changes of 95th percentile of home gait cadence, stride length, stride, stance and swing durations (assessed during 10 days with FeetMe® Insoles) at 12 weeks (MSA subgroup only), 24 and 48 weeks versus baseline | at baseline at 12weeks, at 24 weeks and 48 weeks
Changes of UMSARS I-II versus baseline in MSA subgroup | at baseline at 12weeks, at 24 weeks and 48 weeks
  UMSARS contains four parts, the UMSARS-1 and UMSARS-2 are reported in this outcome. UMSARS-1 scores symptoms of neurological and autonomic dysfunction (12 questions). UMSARS-2 is motor examination (14 questions). All questions range from 0 (normal) to 4(extreme dysfunction). Higher scores mean greater the impairment. Negative change from baseline values indicate improvement.
Changes of MSA-QoL versus baseline in MSA subgroup | at baseline at 24 and 48 weeks
  MSA-QoL is a patient-rated health-related Quality of life scale for patients with multiple system atrophy (MSA). Visual Analog score is designed to determine overall life satisfaction in patient with MSA. Scale is given response option format (0 - extremely unsatisfied with life 100 - extremely satisfied with life), where higher scores indicate better satisfaction/quality of life.
Changes of OHQ versus baseline in MSA subgroup | at baseline at 24 and 48 weeks
  OHQ : Oxford Happiness Questionnaire. The total score ranges from 8 to 54, with a higher number indicating better subjective wellness
Changes of OHSA versus baseline in MSA subgroup | at baseline at 24 and 48 weeks
  Orthostatic Hypotension Symptom Assessment (OHSA) and Orthostatic Hypotension Daily Activities Scale (OHDAS) 10 items measured on a Likert-scale
Changes of BBS versus baseline in MSA subgroup | at baseline at 24 and 48 weeks
  Berg Balance Scale (BBS) is a clinical 14-item scale designed to measure balance
Changes of Modified SE-ADL versus baseline in MSA subgroup | at baseline at 24 and 48 weeks
  The Schwab and England Activities of Daily Living (SE-ADL) evaluates patients' perceptions of global functional capacity and dependence. Scoring is expressed in terms of percentage, in 10 steps from 100 to 0 (100% indicates completely independent, 0% indicates bedridden with impaired vegetative functions), so that the lower the score, the worse the functional status. The assessment is conducted by a trained clinician.
Changes of PDSS-2 versus baseline in MSA subgroup | at baseline at 24 and 48 weeks
  The PDSS-2 is a 15-question instrument designed to simultaneously capture the multidimensional aspects of sleep-related problems and changes in sleep quality.
Changes of COMPASS31 versus baseline in MSA subgroup | at baseline at 24 and 48 weeks
  Composite Autonomic Symptom Score (CONPASS 31) includes 31 questions and it will be used to assess autonomic symptoms that provides clinically relevant scores of autonomic symptom severity based. The higher the score the more autonomic symptoms present
Changes of MOCA versus baseline in MSA subgroup | at baseline at 24 and 48 weeks
MRI changes at 24 and 48 weeks versus baseline. | at baseline at 24 and 48 weeks
  For MSA subgroup and all subgroups
DAT-scan changes at 48 weeks versus baseline. | at baseline at 48 weeks
  For Early PD subgroup
PKG changes at 48 weeks versus baseline | at baseline and at 48 weeks
  in early PD and fluctuating subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Moreau, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France